CLINICAL TRIAL: NCT04492319
Title: The Effect of Addition of Neostigmine to Levobupivacaine in Male Patients Receiving Ultrasound Guided Spermatic Cord Block for Postoperative Analgesia in Testicular Sperm Extraction Surgery:
Brief Title: Addition of Neostigmine to Levobupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-18-2020
Record Dates: First submitted 2020-06-03; First posted 2020-07-30 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Spermatic Cord Block
Keywords: Spermatic Cord Block; Neostigmine; Levobupivacaine
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Drug: Control Test
- neostigmine group (Active Comparator)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Control Test — spermatic cord block by 19 ml Levobupivacaine 0.5% plus 1 ml 0.9 normal saline in each side
  Arms: control group
Drug: Neostigmine — spermatic cord block by 19 ml Levobupivacaine 0.5% plus 1 ml neostigmine 500 μg in each side .
  Arms: neostigmine group

SUMMARY:
Using the spermatic cord block has been of great advantage, as it has been cost saving, efficient technique whether used inon its own or combination with a sedative or . Furthermore, it provides minimal cardiac risks, early case ambulation, satisfactory postoperative pain control, as well as a reduced hospital stay and cost. one of the major drawbacks of spermatic cord block is being a single injection technique, leading to a short postoperative analgesia duration. So, to overcome this flaw some adjuvants were proven to prolong the analgesia duration as neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 to 45 years.
* American Society of Anesthesiologists I-II.
* Undergoing Testicular Sperm Extraction Surgery.
* BMI from 18.5 to 40 kg/m2

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia (bleeding disorders e.g. international normalized ratio >1.5, Prothrombin Concentration <70%, platelet count<100 × 109, use of any anti-coagulants, local infection, etc.).
* Known allergy to local anesthetics.
* ASA III-IV.
* Patients aged less than 18 or more than 60.
* Body mass index >35.:

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — operation in male only
Enrollment: 112 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Time from end of surgery to the first postoperative analgesic request | UP TO 24 HOURE
  (duration of the block).

SECONDARY OUTCOMES:
visual analog scale | UP TO 24 HOURE
  visual analog scale ; 0 is bad / 10: is good
spermatic cord block time | UP TO 1 HOURE
  The mean time needed to perform spermatic cord block
Incidence of complications | up to 24 hours
  complications
Postoperative analgesic use | up to 24 hours
  amount of Acetaminophen used postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Amr wahdan, Principal Investigator — lecture
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
sill working